CLINICAL TRIAL: NCT05213741
Title: Feasibility Trial of Magnetic-assisted Colonoscope Platform
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Principal Investigator, Fat-Moon Suk, Attending physician, Taipei Medical University WanFang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: N202004113
Record Dates: First submitted 2022-01-27; First posted 2022-01-28 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Colonoscopy; Colorectal Cancer
Keywords: Colonoscopy; Magnetic-assisted
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetic-assisted colonoscopy group (Experimental): Participants in this group will recieve magnetic-assisted colonoscopic examination
  Interventions: Device: Autonomous navigation of a magnetic colonoscope

INTERVENTIONS:
Device: Autonomous navigation of a magnetic colonoscope — The proposed magnetic-assisted colonoscope system consists of an megnetic field nevigator, magnetic-assisted colonoscope, and image receiving decoder. All participants will receive the magnetic-assisted colonoscopic examination by using this proposed magnetic-assisted colonoscope system

SUMMARY:
Colorectal cancer (CRC) screening program can reduce colon cancer-related mortality. Current CRC screening methods include stool occult blood and DNA testing, blood based tests and radiologic tests. Colonoscopy is considered the gold standard to detect colorectal neoplasms. Previous studies have estimated that cancer mortality to be 68% to 88% lower among persons who undergo screening colonoscopy than among those who do not. However, colonoscopy is an invasive examination, and 10% to 20% of patients fail to tolerate the procedure; therefore, greatly reduces the success rate of completion of colon examination.

External controllability of capsule endoscope by means of an applied magnetic field is a possible solution to the maneuvering problem. However, there is no effective system with straight forward clinical applicability till now. This is ascribable to a lack of reliable magnetic instrumentation suitable for such a purpose. We have reported that magnetic field navigator (MFN) can effectively control the locomotion of capsule endoscope. We have demonstrated the feasibility and safety of magnetic-assisted capsule endoscope for the examination of upper gastrointestinal tract. In this study, we develop a magnetic-assisted capsule colonoscope by combination of the integrated circuit complementary metal-oxide-semiconductor imaging sensor, light-emitting diode, and magnetic control technology. This magnetic-assisted capsule colonoscope operation system includes a MFN Platform, high-end hand-controlled joystick, combined circuit component, control interface and software. This magnetic-assisted capsule colonoscope operation system creates a friendly operating environment for the operators, and may establishe a novel screening system for the colon.

DETAILED DESCRIPTION:
1. Preparation before examination: All subjects must take bowel cleansing drugs as instructed before magnetically controlled colonoscopy After starting to drink laxatives, subjects should continue their daily activities .
2. Magnetically Controlled Colonoscopy procedure:

   No anesthesia will be used during the magnetically controlled colonoscopy in this experiment.

   The subjects lie down on the magnetic control colonoscopy platform. After the magnetically controlled colonoscopy enters the rectum from the subject's anus, the external magnetron is used to assist and guide the pre-colonoscopy after the magnetically controlled colonoscopy enters the rectum from the subject's anus, and the external magnetron is used to assist and guide the colonoscopy go ahead. During the inspection process, the physician monitors the operation of the magnetically controlled colonoscope throughout the process, and the physician can adjust the movement of the colonoscope when necessary.

   Whole colorectal examination is defined as the colonoscope must be inserted into the ileocecal region, and the cecum must be photographed.
3. Pain assessment during examination:

   During the colonoscopy, the researchers will conduct a questionnaire to the patients to assess the pain..

   The evaluation method is based on the Verbal Scale to evaluate the maximum discomfort, from 0 to 10 points; ; Among them, 0 points are painless, 10 points are the most severe.

   If the patient's pain assessment score is greater than 5 and the patient cannot tolerate colonoscopy, the examination will be terminated.

   If there are difficulties during the examination, and the magnetic-controlled colonoscopy cannot complete the examination within 1 hours, the examination shall be terminated.
4. After the colonoscopy is completed, the researcher conducts an overall pain assessment to the subjects by means of a questionnaire. On the day after the colonoscopy, the researcher asked the subjects whether they would like to accept the next colonoscopy follow-up examination by means of a questionnaire.
5. After the magnetic-controlled colonoscopy, the images and time recorded by the colonoscopy will be interpreted by computer-captured images, and the completion rate of the magnetic-controlled colonoscopy will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

Aged 20-65 health volunteers without any contraindication

Exclusion Criteria:

1. Person allergy to polyethylene glycol.
2. Phenylkentouria
3. Congestive heart failure (NYHA grade 3)
4. Renal function impairment.
5. Difficulty in swallowing, GI perforation, GI bleeding, toxic enterocolitis, toxic colitis, megacolon, diverticulitis, peritonitis
6. Body weight less than 20kg
7. Wrist more than 120cm
8. Gastrointestinal tract obstruction
9. Pregnant woman.
10. Person with electrical medical implantation such as pacemaker, cochlear implant or other medical devices.
11. Person implanted with metal medical device such as metal implantation, metallic stent, metallic denture, metallic valve, metallic joint, metallic joint or plate.
12. Person with history of abdominal surgery.
13. Person with cancer.
14. Person with bleeding tendency
15. Person with asthma
16. History of cardiac infraction, pulmonary embolism, stroke in recent 6 months
17. Heart failure with NYHA grades 4

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of magnetic-assisted colonoscope system | The end of colonoscopic examination
  The completion rate of colonoscopic examination by using the magnetic-assisted colonoscope system
Safety of magnetic-assisted colonoscope system | The end of colonoscopic examination
  The complication rate of colonoscopic examination by using the magnetic-assisted

CONTACTS AND LOCATIONS:
Overall Officials: FAT-MOON SUK, M.D., Principal Investigator — Taipei Medical University Wan Fang Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lien GS, Liu CW, Jiang JA, Chuang CL, Teng MT. Magnetic control system targeted for capsule endoscopic operations in the stomach--design, fabrication, and in vitro and ex vivo evaluations. IEEE Trans Biomed Eng. 2012 Jul;59(7):2068-79. doi: 10.1109/TBME.2012.2198061. Epub 2012 May 7. PMID 22581127
- [Background] Yang CS, Suk FM, Chen CN, Chuang CL, Jiang JA, Liu CW, Lien GS. Colonoscopy with magnetic control system to navigate the forepart of colonoscope shortens the cecal intubation time. Surg Endosc. 2014 Aug;28(8):2480-3. doi: 10.1007/s00464-014-3460-7. Epub 2014 Mar 20. PMID 24648105
- [Background] Huang HE, Yen SY, Chu CF, Suk FM, Lien GS, Liu CW. Autonomous navigation of a magnetic colonoscope using force sensing and a heuristic search algorithm. Sci Rep. 2021 Aug 13;11(1):16491. doi: 10.1038/s41598-021-95760-7. PMID 34389760
- [Background] Lien GS, Wu MS, Chen CN, Liu CW, Suk FM. Feasibility and safety of a novel magnetic-assisted capsule endoscope system in a preliminary examination for upper gastrointestinal tract. Surg Endosc. 2018 Apr;32(4):1937-1944. doi: 10.1007/s00464-017-5887-0. Epub 2017 Oct 25. PMID 29071416
- [Background] Yen SY, Huang HE, Lien GS, Liu CW, Chu CF, Huang WM, Suk FM. Automatic lumen detection and magnetic alignment control for magnetic-assisted capsule colonoscope system optimization. Sci Rep. 2021 Mar 19;11(1):6460. doi: 10.1038/s41598-021-86101-9. PMID 33742067